CLINICAL TRIAL: NCT02993783
Title: An Open-Label, Dose-Finding Study of Vedolizumab IV for Treatment of Steroid-Refractory Acute Intestinal Graft-Versus-Host Disease (GvHD) in Patients Who Have Undergone Allogeneic Hematopoietic Stem Cell Transplantation (Allo-HSCT)
Brief Title: A Dose-Finding Study of Vedolizumab for Treatment of Steroid-Refractory Acute Intestinal Graft-Versus-Host Disease (GvHD) in Participants Who Have Undergone Allogeneic Hematopoietic Stem Cell Transplantation (Allo-HSCT)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of efficacy of the drug; no safety concern
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Vedolizumab-2004; 2016-002985-30 (EudraCT Number); U1111-1185-6832 (Other: WHO)
Record Dates: First submitted 2016-12-08; First posted 2016-12-15 (Estimated); Results first posted 2019-05-24 (Actual); Last update posted 2019-05-24 (Actual); Status verified 2019-05

CONDITIONS: Allogeneic Hematopoietic Stem Cell Transplantation
Keywords: Drug Therapy
MeSH Terms: interventions — vedolizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Vedolizumab 300 mg (Experimental): Vedolizumab 300 mg, intravenous (IV) infusion, once on Days 1, 15, 43, 71 and 99.
  Interventions: Drug: Vedolizumab
- Vedolizumab 600 mg (Experimental): Vedolizumab 600 mg, IV infusion, once on Days 1, 15, 43, 71 and 99.
  Interventions: Drug: Vedolizumab

INTERVENTIONS:
Drug: Vedolizumab — Vedolizumab IV infusion
  Other Names: Entyvio; MLN0002

SUMMARY:
The purpose of this study is to assess the initial activity, tolerability, safety and to identify a recommended dose and regimen of vedolizumab intravenous (IV) administered for treatment of steroid-refractory acute intestinal GvHD in participants who have undergone allo-HSCT.

DETAILED DESCRIPTION:
The drug being tested in this study is called vedolizumab. This study will look at the tolerability and effectiveness of vedolizumab IV in participants with acute intestinal GvHD who have received no systemic therapy for the treatment of acute GvHD (prophylaxis acceptable) other than corticosteroids.

The study enrolled 17 participants. Participants will be randomly assigned (by chance, like flipping a coin) to one of the two treatment groups:

* Vedolizumab 300 mg
* Vedolizumab 600 mg

All participants will be infused intravenously at the same time each day throughout the study. Vedolizumab IV will be administered on Days 1, 15, 43, 71, and 99. After approximately 10 participants are enrolled at each dose level and have data available from the Day 28 evaluation, safety, tolerability, efficacy, and pharmacokinetic (PK), results will be assessed for each dose level, and the appropriate dose for subsequent participants in the study will be determined.

This multi-center trial will be conducted in multiple countries. The overall time to participate in this study is 32 weeks. Participants will make multiple visits to the clinic after last dose of study drug for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Recipient of 1 allogeneic hematopoietic stem cell transplantation (allo-HSCT) but not more than 1 allo-HSCT.
2. Has primary steroid-refractory graft-versus-host disease (GvHD). Steroid-refractory disease is defined as worsening or no improvement in 5 to 7 days of treatment with methylprednisolone 2 milligram per kilogram (mg/kg) or equivalent or lack of a CR after 14 days of primary treatment with methylprednisolone 2 mg/kg or equivalent. Note that participants who develop intestinal GvHD while receiving systemic therapy for other GvHD are still eligible after 5 to 7 days, even if the intestinal GvHD has not been present for the entire duration. Participants who may have received an increase in their steroid dose treatment (example, increased methylprednisolone from 1 mg/kg to 2 mg/kg) before enrollment will be eligible, provided the participant has met the definition of steroid refractory above. Participants who develop toxicity on corticosteroids or who are otherwise medically unable to be dosed to this level, will also be eligible.
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 3.
4. Evidence of myeloid engraftment defined by absolute neutrophil count greater than or equal to (>=) 0.5*109/liter (L) on 3 consecutive days.

Exclusion Criteria:

1. Presence of chronic GvHD at Screening (including acute-chronic overlap syndrome).
2. Relapse of underlying malignant disease after allo-HSCT.
3. Hyperacute GvHD defined as onset of GvHD within the first 15 days following hematopoietic stem cell infusion.
4. Received systemic agents other than corticosteroids for treatment of acute GvHD. GvHD prophylaxis agents (example, calcineurin inhibitors) may be continued.
5. Life expectancy of <3 weeks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2017-04-28 (Actual); Primary Completion 2018-05-09 (Actual); Study Completion 2018-05-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Millennium Pharmaceuticals, Inc.
Locations (15):
- United States (6):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Washington University, St Louis, Missouri
  - Mount Sinai - PRIME, Lake Success, New York
  - OSU - James Comprehensive Cancer Center, Columbus, Ohio
  - Baylor University Medical Center, Dallas, Texas
  - Seattle Cancer Care Alliance, Seattle, Washington
- Belgium (3):
  - ZNA Stuivenberg, Antwerp
  - AZ Sint-Jan Brugge, Bruges
  - UZ Leuven, Leuven
- France (3):
  - CHU Nantes - Hotel Dieu, Nantes, Loire Atlantique
  - Hopital Claude Huriez - CHU Lille, Lille, Nord
  - Hopital Saint-Antoine, Paris, Paris
- Oslo Universitetssykehus - Rikshospitalet, Oslo, Norway
- Sweden (2):
  - Skanes Universitetssjukhus, Lund, Lund
  - Akademiska Sjukhuset, Uppsala

IPD SHARING:
Plan to Share IPD: Yes
Takeda makes patient-level, de-identified data sets and associated documents available after applicable marketing approvals and commercial availability have been received, an opportunity for the primary publication of the research has been allowed, and other criteria have been met as set forth in Takeda's Data Sharing Policy (see www.TakedaClinicalTrials.com/Approach for details). To obtain access, researchers must submit a legitimate academic research proposal for adjudication by an independent review panel, who will review the scientific merit of the research and the requestor's qualifications and conflict of interest that can result in potential bias. Once approved, qualified researchers who sign a data sharing agreement are provided access to these data in a secure research environment.

REFERENCES:
- [Derived] Floisand Y, Schroeder MA, Chevallier P, Selleslag D, Devine S, Renteria AS, Mohty M, Yakoub-Agha I, Chen C, Parfionovas A, Quadri S, Jansson J, Akbari M, Chen YB. A phase 2a randomized clinical trial of intravenous vedolizumab for the treatment of steroid-refractory intestinal acute graft-versus-host disease. Bone Marrow Transplant. 2021 Oct;56(10):2477-2488. doi: 10.1038/s41409-021-01356-0. Epub 2021 Jun 9. PMID 34108672

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 11 investigative sites in the United States, France, Belgium and Norway from 28 April 2017 to 09 May 2018.
Pre-assignment Details: Participants with steroid-refractory acute intestinal graft-versus-host disease (GvHD) who had undergone allogeneic hematopoietic stem cell transplantation (allo-HSCT) were enrolled to receive 300 mg or 600 mg vedolizumab.
Period: Overall Study
Arm/Group | Vedolizumab 300 mg | Vedolizumab 600 mg
Started | 8 | 9
Completed | 2 | 0
Not Completed | 6 | 9
Not completed — Reason not Specified | 6 | 9

BASELINE CHARACTERISTICS:
Population: Safety analysis set (SAS) included all participants who received any amount of the study drug.
Groups:
- Vedolizumab 300 mg: Vedolizumab 300 mg, IV infusion, once on Days 1, 15, 43, 71 and 99.
- Total: Total of all reporting groups
Arm/Group | Vedolizumab 300 mg | Vedolizumab 600 mg | Total
Number analyzed (Participants) | 8 | 9 | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.1 (10.45) | 59.0 (10.87) | 56.7 (10.64)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 4 | 10
  Male | 2 | 5 | 7
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Not Hispanic or Latino | 6 | 9 | 15
  Not Reported | 2 | 0 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 7 | 9 | 16
  Not Reported | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  Belgium | 2 | 2 | 4
  France | 3 | 1 | 4
  Norway | 0 | 1 | 1
  United States | 3 | 5 | 8
Height [Mean (Standard Deviation); unit: cm] — Population: Data for Height is not available for 1 participant from SAS.
  cm
    number analyzed (Participants) | 8 | 8 | 16
    (all) | 170.3 (12.08) | 169.8 (7.87) | 170.0 (9.85)
Weight [Mean (Standard Deviation); unit: kg] | 76.40 (16.900) | 74.01 (22.255) | 75.14 (19.342)
Baseline Eastern Cooperative Oncology Group (ECOG) Status [Count of Participants; unit: Participants] — ECOG assessed participant's performance status on a 6 point scale: 0=Normal activity (fully active, able to carry on all predisease performance without restriction); 1=Symptoms but ambulatory (restricted in physically strenuous activity, but ambulatory and able to carry out work of a light or sedentary nature); 2=In bed <50% of the time (ambulatory and capable of all self-care, but unable to carry out any work activities); 3=In bed >50% of the time (capable of only limited self-care); 4=100% bedridden (completely disabled, cannot carry on any selfcare, totally confined to bed or chair) 5=Dead.
  Participants
    0 | 2 | 0 | 2
    1 | 3 | 2 | 5
    2 | 1 | 4 | 5
    3 | 2 | 3 | 5

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Overall Response (Partial Response [PR]+Very Good Partial Response [VGPR]+Complete Response [CR]) at Day 28
Description: CR is defined as the resolution of all signs and symptoms of acute graft-versus-host-disease (GvHD). VGPR is defined as resolution of the signs and symptoms of the GvHD: 1) Skin: no rash, or residual erythematous rash involving <25% of the body surface, without bullae (excluding residual faint erythema and hyperpigmentation). 2) Liver: total serum bilirubin concentration <2 mg/dL or <25% of baseline at enrollment. 3) Gut: a) participant tolerates food or enteral feeding; b) predominantly formed stools; c) no overt gastrointestinal bleeding or abdominal cramping; d) no more than occasional nausea or vomiting. PR is defined as improvement of 1 GvHD stage in 1 or more organs without progression in any organ.
Time Frame: Day 28
Population: Efficacy analysis set included all participants from the safety set who had baseline efficacy assessment and at least one post-baseline efficacy assessment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Vedolizumab 300 mg | Vedolizumab 600 mg
Number analyzed (Participants) | 8 | 9
percentage of participants | 50.0 [15.7 to 84.3] | 22.2 [2.8 to 60.0]

2. Primary Outcome: Number of Participants Who Experienced Serious Adverse Events (SAEs) Through Day 28
Description: An Adverse Event (AE) is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. An SAE is defined as an untoward medical occurrence, significant hazard, contraindication, side effect or precaution that at any dose: results in death, is life-threatening, required in-patient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect or is medically significant.
Time Frame: From first dose up to Day 28
Population: SAS included all participants who received any amount of the study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Vedolizumab 300 mg | Vedolizumab 600 mg
Number analyzed (Participants) | 8 | 9
Participants | 3 | 4

3. Secondary Outcome: Percentage of Participants Who Died in the Absence of Primary Malignancy Relapse After Allo-HSCT at Month 6
Time Frame: Month 6
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Vedolizumab 300 mg | Vedolizumab 600 mg
Number analyzed (Participants) | 8 | 9
percentage of participants | 50.0 [15.7 to 84.3] | 88.9 [68.4 to 100.0]

4. Secondary Outcome: Percentage of Participants With Acute GvHD Complete Response (CR) at Day 28
Description: CR is defined as the resolution of all signs and symptoms of acute GvHD.
Time Frame: Day 28
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Vedolizumab 300 mg | Vedolizumab 600 mg
Number analyzed (Participants) | 8 | 9
percentage of participants | 12.5 [0.3 to 52.7] | 0 [0 to 0]

5. Secondary Outcome: Percentage of Participants With Intestinal Overall Response at Day 28
Description: Symptoms of acute intestinal GvHD were measured using the BMT CTN-modified International Bone Marrow Transplant Registry Database (IBMTR) index. Intestinal overall response is either CR, VGPR or PR for intestine only. CR is defined as the resolution of all signs and symptoms of GvHD. VGPR is defined as resolution of the majority of signs and symptoms of intestinal GvHD: a) participant tolerates food or enteral feeding; b) predominantly formed stools; c) no overt gastrointestinal bleeding or abdominal cramping; d) no more than occasional nausea or vomiting. PR is defined as improvement of intestinal GvHD by at least 1 stage.
Time Frame: Day 28
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Vedolizumab 300 mg | Vedolizumab 600 mg
Number analyzed (Participants) | 8 | 9
percentage of participants | 62.5 [24.5 to 91.5] | 33.3 [7.5 to 70.1]

6. Secondary Outcome: Kaplan-Meier Estimate of Percentage of Participants Achieving Survival at Months 6 and 12
Description: The Kaplan-Meier estimate reports the percentage of participants surviving at Months 6 and 12.
Time Frame: Months 6 and 12
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Vedolizumab 300 mg | Vedolizumab 600 mg
Number analyzed (Participants) | 8 | 9
percentage of participants
  Month 6 | 0.50 [0.15 to 0.77] | 0.11 [0.01 to 0.39]
  Month 12 | NA [NA to NA] — Percentage and 95% CI was not reached due to low number of participants with events. | NA [NA to NA] — Percentage and 95% CI was not reached due to low number of participants with events.

7. Secondary Outcome: Percentage of Participants Alive Without GvHD or Primary Malignancy Relapse at Months 6 and 12
Time Frame: Months 6 and 12
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Vedolizumab 300 mg | Vedolizumab 600 mg
Number analyzed (Participants) | 8 | 9
percentage of participants
  Month 6 | 37.5 | 0
  Month 12 | 0 | 0

8. Secondary Outcome: Total Dose of Steroids Administered
Description: Total Steroids administered in mg/kg/day of methylprednisolone or equivalent
Time Frame: From first dose of study drug up to Months 6 and 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/kg/day
Arm/Group | Vedolizumab 300 mg | Vedolizumab 600 mg
Number analyzed (Participants) | 8 | 9
mg/kg/day
  Month 6 | 0.862 (0.6397) | 0.876 (0.4796)
  Month 12 | 0.829 (0.6611) | 0.876 (0.4798)

9. Secondary Outcome: Number of Participants Who Experienced Treatment Emergent Adverse Events (TEAEs)
Description: An AE is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (example, a clinically significant abnormal laboratory finding), symptom, or disease temporally associated with the use of a drug, whether or not it is considered related to the drug. A TEAE is defined as an adverse event with an onset that occurs after receiving study drug.
Time Frame: From first dose of study drug to 18 weeks after last dose (Up to Week 32)
Population: SAS included all participants who received any amount of the study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Vedolizumab 300 mg | Vedolizumab 600 mg
Number analyzed (Participants) | 8 | 9
Participants | 8 | 9

10. Secondary Outcome: Number of Participants Who Experienced Serious Adverse Events (SAEs) Through Week 32
Description: An AE is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. An SAE is defined as an untoward medical occurrence, significant hazard, contraindication, side effect or precaution that at any dose: results in death, is life-threatening, required in-patient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect or is medically significant.
Time Frame: From first dose of study drug to 18 weeks after last dose (Up to Week 32)
Population: SAS included all participants who received any amount of the study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Vedolizumab 300 mg | Vedolizumab 600 mg
Number analyzed (Participants) | 8 | 9
Participants | 6 | 9

11. Secondary Outcome: Number of Participants With Markedly Abnormal Laboratory Parameters Values
Description: Clinical Laboratory parameters included tests for chemistry, hematology and urinalysis. Markedly abnormal values during treatment period were categorized as:alanine aminotransferase (ALT)>3.0 U/L*upper limit of normal(ULN),albumin<25 g/L*lower limit of normal(LLN),alkaline phosphatase >3.0 U/L*ULN,aspartate aminotransferase >3.0 U/L*ULN,bilirubin >2 umol/L*ULN,blood urea nitrogen(BUN) >10.7 mmol/L,calcium <1.75 mmol/L, >2.88 mmol/L,chloride <75 mmol/L, >126 mmol/L,creatinine >177umol/L,gamma glutamyl transferase (GGT) >3 U/L*ULN,glucose <2.8 mmol/L, >19.4 mmol/L,phosphate <0.52 mmol/L, >2.10 mmol/L,potassium<3 mmol/L, >6 mmol/L,sodium <130 mmol/L, >150 mmol/L,basophils >3(10^9/L)*ULN,eosinophils >2(10^9/L)*ULN,hematocrit (%) <0.8*LLN, >1.2*ULN,hemoglobin <0.8 g/L*LLN, >1.2 g/L*ULN,leukocytes <0.5 (10^9/L)*LLN, >1.5 (10^9/L)*ULN,lymphocytes <0.5 (10^9/L)*LLN, >1.5(10^9/L)*ULN,monocytes >2 (10^9/L)*ULN,neutrophils <0.5(10^9/L)*LLN, >1.5 (10^9/L)*ULN,platelets <75(10^9/L), >600(10^9/L).
Time Frame: From Baseline up to last dose of study drug (Day 99)
Population: SAS included all participants who received any amount of the study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Vedolizumab 300 mg | Vedolizumab 600 mg
Number analyzed (Participants) | 8 | 9
Participants
  ALT >3.0 U/L*ULN | 4 | 0
  Albumin <25 g/L*LLN | 4 | 8
  Alkaline phosphatase >3.0 U/L*ULN | 1 | 0
  Aspartate aminotransferase >3.0 U/L*ULN | 1 | 0
  Bilirubin >2 umol/L*ULN | 1 | 2
  BUN >10.7 mmol/L | 3 | 6
  Calcium <1.75 mmol/L | 0 | 3
  Calcium >2.88 mmol/L | 0 | 0
  Chloride <75 mmol/L | 0 | 0
  Chloride >126 mmol/L | 0 | 0
  Creatinine >177umol/L | 0 | 1
  GGT >3 U/L*ULN | 5 | 2
  Glucose <2.8 mmol/L | 0 | 0
  Glucose >19.4 mmol/L | 1 | 0
  Phosphate <0.52 mmol/L | 0 | 0
  Phosphate >2.10 mmol/L | 0 | 1
  Potassium <3 mmol/L | 1 | 0
  Potassium >6 mmol/L | 0 | 0
  Sodium <130 mmol/L | 0 | 0
  Sodium >150 mmol/L | 0 | 0
  Basophils >3(10^9/L)*ULN | 0 | 0
  Eosinophils >2(10^9/L)*ULN | 0 | 0
  Hematocrit (%) <0.8*LLN | 7 | 8
  Hematocrit (%) >1.2*ULN | 0 | 0
  Hemoglobin <0.8 g/L*LLN | 7 | 8
  Hemoglobin >1.2 g/L*ULN | 0 | 0
  Leukocytes <0.5 (10^9/L)*LLN | 3 | 7
  Leukocytes >1.5 (10^9/L)*ULN | 1 | 0
  Lymphocytes <0.5 (10^9/L)*LLN | 7 | 9
  Lymphocytes >1.5(10^9/L)*ULN | 0 | 0
  Monocytes >2 (10^9/L)*ULN | 0 | 1
  Neutrophils <0.5(10^9/L)*LLN | 0 | 3
  Neutrophils >1.5 (10^9/L)*ULN | 1 | 1
  Platelets <75(10^9/L) | 8 | 9
  Platelets >600(10^9/L) | 0 | 0

12. Secondary Outcome: Number of Participants With Markedly Abnormal Vital Signs
Description: Vital signs included heart rate, respiratory rate, systolic and diastolic blood pressure, temperature and weight. The vital sign values outside the range: systolic blood pressure (SBP) <85 mmHg and change from Baseline (BL) <=-20 mmHg, >180 mmHg and change from Baseline >=20 mmHg,diastolic blood pressure (DBP) <50 mmHg and change from Baseline <=-15 mmHg, >110 mmHg and change from Baseline >=15 mmHg, heart rate <50 beats per minute (bpm),>120 beats per minute, temperature <35.6 Degree C, >37.7 Degree C and weight change from Baseline <=-7 % and weight change from Baseline >=7 % assessed during treatment period were considered markedly abnormal.
Time Frame: From Baseline up to last dose of study drug (Day 99)
Population: SAS included all participants who received any amount of the study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Vedolizumab 300 mg | Vedolizumab 600 mg
Number analyzed (Participants) | 8 | 9
Participants
  SBP <85 mmHg and change from BL <=-20 mmHg | 0 | 0
  SBP >180 mmHg and change from BL >=20 mmHg | 1 | 0
  DBP <50 mmHg and change from BL<=-15 mmHg | 0 | 0
  DBP >110 mmHg and change from BL>=15 mmHg | 0 | 0
  Heart Rate <50 bpm | 0 | 0
  Heart Rate >120 bpm | 0 | 1
  Temperature <35.6 Degree C | 1 | 3
  Temperature >37.7 Degree C | 0 | 0
  Weight change from BL <=-7 % | 4 | 2
  Weight change from BL >=7 % | 3 | 1

13. Secondary Outcome: Ctrough: Trough Serum Concentrations of Vedolizumab
Time Frame: Day 99 (pre-dose)
Population: Pharmacokinetic (PK) set included all participants from the safety set with at least 1 post dose PK sample collected.
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Vedolizumab 300 mg | Vedolizumab 600 mg
Number analyzed (Participants) | 8 | 8
ug/mL | 40.2 (37.2) | 12.3 (5.49)

ADVERSE EVENTS:
Time Frame: From first dose of study drug to 18 weeks after the last dose of study drug (Up to approximately 32 weeks)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Vedolizumab 300 mg | Vedolizumab 600 mg
All-Cause Mortality (participants affected / at risk) | 4/8 | 9/9
Serious Adverse Events (participants affected / at risk) | 6/8 | 9/9
Other Adverse Events (participants affected / at risk) | 8/8 | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vedolizumab 300 mg (N=8) | Vedolizumab 600 mg (N=9)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 1
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Death (General disorders) | 1 | 0
Graft versus host disease (Immune system disorders) | 0 | 3
Acute graft versus host disease (Immune system disorders) | 0 | 1
Acute graft versus host disease in intestine (Immune system disorders) | 1 | 0
Acute graft versus host disease in liver (Immune system disorders) | 0 | 1
Graft versus host disease in gastrointestinal tract (Immune system disorders) | 0 | 1
Peritonitis (Infections and infestations) | 0 | 1
Bacterial sepsis (Infections and infestations) | 1 | 0
Citrobacter sepsis (Infections and infestations) | 0 | 1
Cytomegalovirus colitis (Infections and infestations) | 0 | 1
Enterococcal sepsis (Infections and infestations) | 1 | 1
Escherichia infection (Infections and infestations) | 0 | 1
Mediastinitis (Infections and infestations) | 0 | 1
Pneumonia necrotising (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 2 | 1
Urosepsis (Infections and infestations) | 1 | 0
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Tremor (Nervous system disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 1
Haematoma (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vedolizumab 300 mg (N=8) | Vedolizumab 600 mg (N=9)
Anaemia (Blood and lymphatic system disorders) | 4 | 3
Neutropenia (Blood and lymphatic system disorders) | 1 | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 1
Aplasia pure red cell (Blood and lymphatic system disorders) | 1 | 0
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Pericardial effusion (Cardiac disorders) | 1 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 1
Adrenal insufficiency (Endocrine disorders) | 0 | 1
Vision blurred (Eye disorders) | 2 | 0
Dry eye (Eye disorders) | 0 | 1
Eye pruritus (Eye disorders) | 0 | 1
Lacrimation increased (Eye disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 2
Nausea (Gastrointestinal disorders) | 3 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 1
Vomiting (Gastrointestinal disorders) | 2 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Ascites (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 1
Gingival pain (Gastrointestinal disorders) | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0
Ileus paralytic (Gastrointestinal disorders) | 1 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Mouth ulceration (Gastrointestinal disorders) | 1 | 0
Oral mucosa haematoma (Gastrointestinal disorders) | 1 | 0
Proctalgia (Gastrointestinal disorders) | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1
Stomatitis (Gastrointestinal disorders) | 1 | 0
Tongue discolouration (Gastrointestinal disorders) | 0 | 1
Oedema peripheral (General disorders) | 3 | 3
Fatigue (General disorders) | 0 | 3
Pyrexia (General disorders) | 1 | 2
Generalised oedema (General disorders) | 1 | 1
Asthenia (General disorders) | 1 | 0
Catheter site haemorrhage (General disorders) | 0 | 1
Chills (General disorders) | 1 | 0
Injection site pain (General disorders) | 1 | 0
Oedema (General disorders) | 1 | 0
Pain (General disorders) | 1 | 0
Hypogammaglobulinaemia (Immune system disorders) | 2 | 1
Graft versus host disease in gastrointestinal tract (Immune system disorders) | 0 | 2
Graft versus host disease in skin (Immune system disorders) | 1 | 1
Acute graft versus host disease in intestine (Immune system disorders) | 1 | 0
Acute graft versus host disease in skin (Immune system disorders) | 1 | 0
Cytomegalovirus infection (Infections and infestations) | 2 | 1
BK virus infection (Infections and infestations) | 1 | 1
Enterococcal infection (Infections and infestations) | 1 | 1
Klebsiella infection (Infections and infestations) | 1 | 1
Staphylococcal infection (Infections and infestations) | 0 | 2
Urinary tract infection enterococcal (Infections and infestations) | 1 | 1
Aspergillus infection (Infections and infestations) | 0 | 1
Clostridial infection (Infections and infestations) | 1 | 0
Clostridium difficile infection (Infections and infestations) | 1 | 0
Corona virus infection (Infections and infestations) | 1 | 0
Cytomegalovirus colitis (Infections and infestations) | 1 | 0
Device related infection (Infections and infestations) | 0 | 1
Enterobacter infection (Infections and infestations) | 1 | 0
Escherichia infection (Infections and infestations) | 0 | 1
Escherichia urinary tract infection (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 0 | 1
Mastoiditis (Infections and infestations) | 0 | 1
Otitis externa (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1
Pseudomonas infection (Infections and infestations) | 0 | 1
Septic shock (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1
Urinary tract infection bacterial (Infections and infestations) | 1 | 0
Urosepsis (Infections and infestations) | 1 | 0
Vaginal infection (Infections and infestations) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 1 | 0
Blood bilirubin increased (Investigations) | 2 | 2
Gamma-glutamyltransferase increased (Investigations) | 1 | 2
Platelet count decreased (Investigations) | 2 | 1
White blood cell count decreased (Investigations) | 1 | 2
Alanine aminotransferase increased (Investigations) | 1 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 1
Blood alkaline phosphatase increased (Investigations) | 1 | 1
Blood urea increased (Investigations) | 0 | 2
BK polyomavirus test positive (Investigations) | 0 | 1
Blood beta-D-glucan increased (Investigations) | 0 | 1
Blood creatine increased (Investigations) | 0 | 1
Blood pressure decreased (Investigations) | 0 | 1
Cytomegalovirus test positive (Investigations) | 0 | 1
Electrocardiogram QT prolonged (Investigations) | 0 | 1
Liver function test abnormal (Investigations) | 1 | 0
Neutrophil count decreased (Investigations) | 0 | 1
Oxygen saturation decreased (Investigations) | 0 | 1
Urine output decreased (Investigations) | 0 | 1
Vitamin D decreased (Investigations) | 0 | 1
Weight decreased (Investigations) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 5
Hyperglycaemia (Metabolism and nutrition disorders) | 3 | 2
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 | 3
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 3
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 2
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 | 2
Acidosis (Metabolism and nutrition disorders) | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 1
Fluid imbalance (Metabolism and nutrition disorders) | 0 | 1
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1
Malnutrition (Metabolism and nutrition disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 3
Headache (Nervous system disorders) | 1 | 1
Somnolence (Nervous system disorders) | 0 | 2
Ageusia (Nervous system disorders) | 0 | 1
Clonus (Nervous system disorders) | 0 | 1
Embolic stroke (Nervous system disorders) | 0 | 1
Head titubation (Nervous system disorders) | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 0
Paraesthesia (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 0 | 1
Tremor (Nervous system disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 1
Anxiety (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 1
Pollakiuria (Renal and urinary disorders) | 0 | 1
Proteinuria (Renal and urinary disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 1
Oedema genital (Reproductive system and breast disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Increased bronchial secretion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pain of skin (Skin and subcutaneous tissue disorders) | 1 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 0
Blister (Skin and subcutaneous tissue disorders) | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1 | 0
Lichen planus (Skin and subcutaneous tissue disorders) | 1 | 0
Onychoclasis (Skin and subcutaneous tissue disorders) | 0 | 1
Rash macular (Skin and subcutaneous tissue disorders) | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1
Hypotension (Vascular disorders) | 1 | 2
Haematoma (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 1
Jugular vein thrombosis (Vascular disorders) | 0 | 1
Venoocclusive disease (Vascular disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-09-13): https://cdn.clinicaltrials.gov/large-docs/83/NCT02993783/SAP_000.pdf
  • Study Protocol (2017-11-27): https://cdn.clinicaltrials.gov/large-docs/83/NCT02993783/Prot_001.pdf